CLINICAL TRIAL: NCT02775890
Title: A Prospective Observational Cohort Study Assessing the Feasibility of Measuring Serum Lead Levels in New Zealand Hunters Using Lead Projectiles
Brief Title: Potential Lead Exposure Through Eating Self-harvested Wild Game
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nelson Marlborough Institute of Technology (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1NMIT2016
Record Dates: First submitted 2016-05-10; First posted 2016-05-18 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Lead; Toxicology

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eating lead-shot wild game: Hunters that have eaten lead-shot in the past week will have blood lead levels measured.
  Interventions: Behavioral: Eating wild game shot with lead bullets
- Not eating lead-shot wild game: Hunters that have not eaten lead-shot in the past week will have blood lead levels measured.

INTERVENTIONS:
Behavioral: Eating wild game shot with lead bullets — Participants will eat meat harvested with lead bullets, prepare mince meat and eat at least a standard serving (>85 grams).
  Groups: Eating lead-shot wild game

SUMMARY:
This is a clinical research protocol to determine the feasibility of assessing lead levels in hunters who use lead projectiles. This study will determine if it is possible to perform an interventional double-blind placebo-controlled study of lead levels in hunters using lead or lead-free projectiles following consumption of self-harvested wild game. The hypothesis for the subsequent study is that minute lead particles from shrapnel dispersed through the animal during harvest are ingested and result in increased lead serum levels. This current observational study establishes if this conclusive interventional study is possible through establishing if hunters using lead projectiles in New Zealand have elevated lead levels after eating animals harvested with lead projectiles. This study will be conducted in compliance with the protocol, Good Clinical Practice Standards, associated regulations and institutional research requirements.

This study aims to assess if hunters eating meat shot with lead projectiles experience elevated lead levels. Hunters will be asked to provide blood samples 2-4 days after they eat meat harvested with lead bullets and provide a subsequent sample when they have abstained from eating wild game harvested with lead bullets. We have chosen to use deer as the species for this study to reduce variation and New Zealand is the ideal place to conduct this study because of year-round hunting of deer. This design will allows paired testing of subject lead levels.

ELIGIBILITY:
Inclusion Criteria:

* New Zealand firearms license

Exclusion Criteria:

* Smoker
* Any type of kidney dysfunction
* Individuals working in the following industries that may entail lead exposure:

  1. lead-acid battery manufacture
  2. lead smelting
  3. non-ferrous smelting and casting (e.g. brass)
  4. steel scrap smelting
  5. scrap lead metal handling
  6. cutting/welding steel scrap
  7. machining or polishing lead-containing alloys
  8. plastic production (where lead compounds are used as stabilisers)
  9. demolition
  10. lead soldering
  11. plastic recycling
  12. panel beating
  13. paint removal
  14. sandblasting
  15. leadlight window manufacture
  16. lead casting, e.g. fishing weights, toy soldiers
  17. radiator repair,
  18. car exhaust repair and engine reconditioning (for older makes and models of vehicles)
  19. jewellery (silver) production
  20. shooting range

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hunters eating self-harvested wild game with lead bullets.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Lead levels | Within one year, after participants have eaten a meal (>85grams) of lead-shot meat
  A paired t-test will be conducted comparing lead levels in participants when eating wild game harvested with lead projectiles and when participants have not eaten wild game harvested with lead projectiles.

SECONDARY OUTCOMES:
Complete blood cell counts | Within one year, after participants have eaten a meal (>85grams) of lead-shot meat
  Paired-t tests comparing data from the complete blood count will be performed
Correlation between lead levels and complete blood cell counts | At close of study, within one year
Correlation between lead bullet mass and blood lead levels | At close of study, within one year

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Buenz, PhD, Principal Investigator — Nelson Marlborough Institute of Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buenz EJ. Lead Exposure Through Eating Wild Game. Am J Med. 2016 May;129(5):457-8. doi: 10.1016/j.amjmed.2015.12.022. Epub 2016 Jan 18. No abstract available. PMID 26797078
- [Background] Buenz EJ. Eliminating potential lead exposure in imported New Zealand wild game. Public Health. 2016 Oct;139:236-237. doi: 10.1016/j.puhe.2016.06.025. Epub 2016 Jul 22. No abstract available. PMID 27456932
- [Background] Buenz EJ, Parry GJ, Peacey M. Consumption of wild-harvested meat from New Zealand feral animals provides a unique opportunity to study the health effects of lead exposure in hunters. Ambio. 2016 Sep;45(5):629-31. doi: 10.1007/s13280-016-0798-1. Epub 2016 Jun 25. No abstract available. PMID 27344321
- [Background] Buenz EJ. Non-lead ammunition may reduce lead levels in wild game. Environ Sci Pollut Res Int. 2016 Aug;23(15):15773. doi: 10.1007/s11356-016-7020-7. Epub 2016 Jun 8. No abstract available. PMID 27272923
- [Derived] Buenz EJ, Parry GJ, Bauer BA, Matheny LM, Breukel K. A prospective observational study assessing the feasibility of measuring blood lead levels in New Zealand hunters eating meat harvested with lead projectiles. Contemp Clin Trials Commun. 2017 Feb 8;5:137-143. doi: 10.1016/j.conctc.2017.02.002. eCollection 2017 Mar. PMID 29740629